CLINICAL TRIAL: NCT02649842
Title: Post-Approval Study of the TECNIS® Toric IOL Extended Cylinder Range (ECR), Models ZCT450, ZCT525 and ZCT600
Brief Title: Post-Approval Study of the TECNIS® Toric Extended Cylinder Range Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Optics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TIOL-204-EPAS
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Cataract; Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Extended Cylinder IOL (Experimental): Approved toric intraocular lenses, Model ZCT450, ZCT525 or ZCT600
  Interventions: Device: TECNIS Toric Models ZCT450, ZCT525 or ZCT600

INTERVENTIONS:
Device: TECNIS Toric Models ZCT450, ZCT525 or ZCT600 — Approved toric intraocular lens

SUMMARY:
This study is a prospective, multicenter, bilateral, non-randomized, open-label, clinical study conducted at up to 20 sites in the USA. Subjects were to be bilaterally implanted with one eye having an extended cylinder (high cylinder) toric IOL (model ZCT450, ZCT525 or ZCT600) and the fellow eye having a high cylinder toric IOL (model ZCT450, ZCT525 or ZCT600) or a lower cylinder toric IOL (ZCT300 or ZCT400). This study evaluates the outcomes for subjects implanted with at least one higher cylinder toric IOL.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the performance of the higher cylinder (ZCT450,ZCT525 and ZCT600) toric IOLs. Some subjects had the higher cylinder toric IOLs in both eyes with other subjects having a higher cylinder toric IOL in one eye and the lower cylinder toric IOL in the other eye.

Per the statistical plan, data for the ZCT450/525/600 toric IOLs were to be pooled together and reported as one group.

The primary endpoint is the rate of severe visual distortions reported by subject at 6 months via questionnaire. The analysis population for this endpoint will be bilaterally implanted subjects with a high cylinder IOL (ZCT450/525/600) in the primary eye and a high cylinder IOL (ZCT450/525/600) or a low cylinder IOL (ZCT300/400) in the fellow eye.

There were no formal secondary endpoints. Data from a few other endpoints (rate of IOL repositioning due to IOL misalignment and percent change in cylinder) have been reported. For these endpoints the analysis population contains all subjects implanted with a ZCT450/525/600 in at least one eye.

Adverse events were reported by subject for all subjects with a high cylinder IOL (ZCT450/525/600) in at least one eye.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 22 years of age
* Bilateral cataracts
* Preoperative keratometric cylinder of at least 2.00 D in both eyes with at least one eye having approximately 3.00 D to 4.75 D of corneal astigmatism.
* Ability to understand, read and write English in order to consent to study participation and complete a study questionnaire
* Signed informed consent and HIPAA authorization

Exclusion Criteria:

* Irregular corneal astigmatism
* Any corneal pathology/abnormality other than regular corneal astigmatism
* Previous corneal surgery or recent ocular trauma or intraocular surgery that is not resolved/stable or may affect visual outcomes
* Any pupil abnormalities
* Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration
* Known ocular disease or pathology that may affect visual acuity or that may require surgical intervention during the course of the study
* Concurrent participation or participation during 30 days prior to preoperative visit in any other clinical study
* Planned monovision correction
* Patient is pregnant, plans to become pregnant or is lactating

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-03-21 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Devi Priya Janakiraman, OD,FAAO, Study Director — Abbott Medical Optics

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per SAP there is only one arm. It includes all subjects with ZCT450/525/600 toric IOL in the primary eye.Fellow eye can have the same IOL or a ZCT300/400.
Groups:
- Extended Cylinder IOL: All subjects implanted with an extended cylinder IOL (ZCT450, ZCT525 or ZCT600) in at least one eye.
Period: Overall Study
Arm/Group | Extended Cylinder IOL
Started | 101
Completed | 101
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All subjects with an extended (high) cylinder IOL (ZCT450, ZCT525 or ZCT600) in at least one eye.Per the statistical plan, data for the ZCT450,ZCT525 and ZCT600 toric IOLs were to be pooled together and reported as one group.
Units Other Than Participants: Primary Eyes
Arm/Group | Extended Cylinder IOL
Number analyzed (Participants) | 101
Number analyzed (Primary Eyes) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 94
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Rate of Severe Visual Distortions
Description: Rate of severe visual distortions based on data from a self administered subject questionnaire
Time Frame: 6 months
Population: All subjects implanted with a high cylinder toric IOL (model ZCT450, ZCT525 or ZCT600) in at least one eye and a high cylinder or low cylinder toric IOL in the fellow eye.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Cylinder IOL
Number analyzed (Participants) | 100
Participants | 3

2. Other Pre Specified Outcome: Rate of IOL Repositioning Due to IOL Misalignment
Description: Rate of IOL repositioning due to IOL misalignment in primary and fellow eyes with a high cylinder toric IOL
Time Frame: 6 months
Population: All subjects implanted with a ZCT450/525/600 in at least one eye
Measure: Count of Participants; unit: Participants
Groups:
- Extended Cylinder IOL: All subjects implanted with an extended cylinder IOL (ZCT450, ZCT525 or ZCT600)
Arm/Group | Extended Cylinder IOL
Number analyzed (Participants) | 101
Participants | 11

3. Other Pre Specified Outcome: Percent Change in Cylinder
Description: Percent change in cylinder= ((postop refractive cylinder-preop keratometric cylinder) / (Target refractive cylinder-preop keratometric cylinder))*100
Time Frame: 6 months
Population: All subjects implanted with a ZCT450/525/600 in at least one eye
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Extended Cylinder IOL: All subjects implanted with a ZCT450/525/600 in at least one eye
Arm/Group | Extended Cylinder IOL
Number analyzed (Participants) | 101
Percent change | 88.36 (21.09)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Extended Cylinder IOL: All subjects implanted with an extended cylinder IOL (ZCT450, ZCT525 or ZCT600) in at least one eye. Subject is considered to have adverse events whether the adverse event was in the higher cylinder or lower cylinder group.
Arm/Group | Extended Cylinder IOL
All-Cause Mortality (participants affected / at risk) | 0/101
Serious Adverse Events (participants affected / at risk) | 19/101
Other Adverse Events (participants affected / at risk) | 1/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Cylinder IOL (N=101)
Lens misalignment requiring IOL repositioning (Surgical and medical procedures) | 11 (12) — 6 participants (6 events) with ZCT600, 4 participants (5 events) with ZCT450 and 1 participant (1 event) with ZCT400
Hyphema (Eye disorders) | 1 (1) — 1 participant implanted with ZCT400
Cystoid Macular Edema (Eye disorders) | 1 (1) — 1 participant implanted with ZCT525
Hospitalization due to fall and broken hip (Injury, poisoning and procedural complications) | 1 (1)
Squamous Cell Carcinoma - Left second finger (Skin and subcutaneous tissue disorders) | 1 (1)
Hospitalization due to unsteady gait/dizziness (General disorders) | 1 (1)
Hospitalization due to appendectomy due to appendicitis (Surgical and medical procedures) | 1 (1)
Hospitalization due to motorcycle accident (Injury, poisoning and procedural complications) | 1 (1)
Lens exchange due to residual astigmatism and myopia (Surgical and medical procedures) | 1 (1) — 1 participant implanted with ZCT525
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extended Cylinder IOL (N=101)
Iridocyclitis (Eye disorders) | 1 (1) — 1 participant implanted with ZCT450

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review results communication prior to public release and can embargo communications regarding trial results at any time.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT02649842/Prot_000.pdf
  • Statistical Analysis Plan (2015-05-29): https://cdn.clinicaltrials.gov/large-docs/42/NCT02649842/SAP_001.pdf